CLINICAL TRIAL: NCT02511249
Title: Early Determinants of Multidimensional Outcome at School Age After Neonatal Arterial Ischemic Stroke (AVCnn7 Years Study)
Brief Title: Early Determinants of Multidimensional Outcome at School Age After Neonatal Arterial Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government); University Hospital of Saint-Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1008026; ANSM (Other: 2010-A00329-30)
Record Dates: First submitted 2015-07-24; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Cerebral Infarction
Keywords: neonatal arterial ischemic stroke; language development; global intellectual functioning; motor abilities
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cohort: 1 evaluation day : The evaluation team included a neuropsychologist, a speech therapist and either a pediatric neurologist or a pediatric physical and rehabilitation medicine practitioner.
  tests carried out : Global intellectual functioning (WISC-IV), Oral language (N-EEL), Gross and fine motor abilities (clinical examination, Box & Block test, 9 Hole Peg test)

SUMMARY:
While perinatal ischemic stroke is the most frequent form of childhood stroke, early determinants of outcome remain poorly understood. Two main structural biases limit the accuracy of most studies: heterogeneity of the population and short follow-up.

Perinatal ischemic stroke includes several conditions that differ in pathophysiology and timing of occurrence. Yet, it is not surprising that risk factors and outcome depend primarily on the type of stroke. Age at evaluation also plays a major role after a neonatal insult. Even though the original lesion is static and focal in perinatal stroke, its consequences grow over time within the maturing brain and affect all fields of neurodevelopment.

The objective of the AVCnn study was to delineate the determinants, clinical and imaging presentation, mechanism, and long term outcome of a category of perinatal stroke (neonatal arterial ischemic stroke: NAIS). This led to the AVCnn cohort, which now gives us the opportunity to regularly monitor a large cohort of children having suffered an NAIS.

DETAILED DESCRIPTION:
Between November 2003 and October 2006, a cohort of one hundred symptomatic term newborns with AIS confirmed through early brain imaging has been constituted.

Regular contacts with the families and their local physician have been maintained since enrollment. In 2010, families were asked through postal mail to participate in the 7 years assessment (AVCnn7ans). Those who accepted were contacted by phone by the coordinators of the study during the months preceding the child's seventh birthday and invited to attend a presentation in person of the current project. This evaluation took place face-to-face for a whole day in a medical setting close to the family residence. The evaluation team included a neuropsychologist, a speech therapist and either a pediatric neurologist or a pediatric physical and rehabilitation medicine practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Belonging to the AVCnn cohort

Exclusion Criteria:

* Lost to follow-up at 7 years.
* Refusal to participate in the current assessment.

Ages: 7 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who have had an ischemic arterial stroke between November 2003 and October 2006, in France, who was included in "AVCnn cohort" and who accept an psychological and physical examination at 7 years
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Epileptic outcome | at 7 years
  Occurrence of two or more afebrile unprovoked seizures after the neonatal period or, in the event of single afebrile unprovoked seizure, when it was decided to introduce antiepileptic treatment
Academic outcome (composite measure) | at 7 years
  Grade retention or the need for specific and individualized support in mainstream school or inclusion in a special school.
Neurodevelopmental outcome at 7 years | at 7 years
  permanent abnormal tone or decreased strength associated with a patent functional deficit

SECONDARY OUTCOMES:
Cerebral imaging ancillary study | at 7 years
  Anatomic post-lesional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane CHABRIER, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (5):
- France (5):
  - Chu D'Angers, Angers
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Chu de Brest, Brest
  - Hopital Necker, Paris
  - Chu de Saint Etienne, Saint-Etienne

REFERENCES:
- [Derived] Thebault G, Martin S, Brouillet D, Brunel L, Dinomais M, Presles E, Fluss J, Chabrier S; AVCnn Study Group. Manual dexterity, but not cerebral palsy, predicts cognitive functioning after neonatal stroke. Dev Med Child Neurol. 2018 Oct;60(10):1045-1051. doi: 10.1111/dmcn.13752. Epub 2018 Apr 6. PMID 29624666
- [Derived] Dinomais M, Thebault G, Hertz-Pannier L, Gautheron V, Nguyen The Tich S, Fluss J, Chabrier S; AVCnn Study Group. Is there an excess of left-handedness after neonatal stroke? Cortex. 2017 Nov;96:161-164. doi: 10.1016/j.cortex.2017.08.007. Epub 2017 Aug 16. No abstract available. PMID 28893386
- [Derived] Groeschel S, Hertz-Pannier L, Delion M, Loustau S, Husson B, Kossorotoff M, Renaud C, Nguyen The Tich S, Chabrier S, Dinomais M; AVCnn study group. Association of transcallosal motor fibres with function of both hands after unilateral neonatal arterial ischemic stroke. Dev Med Child Neurol. 2017 Oct;59(10):1042-1048. doi: 10.1111/dmcn.13517. Epub 2017 Aug 17. PMID 28815625
- [Derived] Dinomais M, Hertz-Pannier L, Groeschel S, Delion M, Husson B, Kossorotoff M, Renaud C, Chabrier S, The Tich SN; AVCnn Study Group. Does Contralesional Hand Function After Neonatal Stroke Only Depend on Lesion Characteristics? Stroke. 2016 Jun;47(6):1647-50. doi: 10.1161/STROKEAHA.116.013545. Epub 2016 May 10. PMID 27165960
- [Derived] Chabrier S, Peyric E, Drutel L, Deron J, Kossorotoff M, Dinomais M, Lazaro L, Lefranc J, Thebault G, Dray G, Fluss J, Renaud C, Nguyen The Tich S; Accident Vasculaire Cerebral du nouveau-ne (AVCnn; [Neonatal Stroke]) Study Group. Multimodal Outcome at 7 Years of Age after Neonatal Arterial Ischemic Stroke. J Pediatr. 2016 May;172:156-161.e3. doi: 10.1016/j.jpeds.2016.01.069. Epub 2016 Mar 9. PMID 26968833